CLINICAL TRIAL: NCT00774267
Title: Evaluation Of Changes In Mammographic Breast Density Associated With Bazedoxifene Acetate/Conjugated Estrogens, Raloxifene And Placebo In Postmenopausal Women: An Ancillary Study Of Protocol 3115A1-303-WW
Brief Title: Study Evaluating Changes In Mammographic Breast Density
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3115A1-4000; B2311010
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1
  Interventions: Drug: BZA 20 mg/CE 0.45 mg
- 2
  Interventions: Drug: BZA 20 mg/CE 0.625 mg
- 3
  Interventions: Drug: Raloxifene 60 mg
- 4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BZA 20 mg/CE 0.45 mg — There was no drug taken during study 3115A1-4000. During the 3115A1-303 study the test article was supplied as baxedoxifene/CE tablets in capsules. Subjects took one capsule orally, once daily at approximately the same time each day on a continuous regimen for 2 years or until early termination from the study.
  Groups: 1
Drug: BZA 20 mg/CE 0.625 mg — There was no drug taken during study 3115A1-4000. During the 3115A1-303 study the test article was supplied as baxedoxifene/CE tablets in capsules. Subjects took one capsule orally, once daily at approximately the same time each day on a continuous regimen for 2 years or until early termination from the study.
  Groups: 2
Drug: Raloxifene 60 mg — There was no drug taken during study 3115A1-4000. During the 3115A1-303 study the test article was supplied as raloxifene tablets in capsules. Subjects took one capsule orally, once daily at approximately the same time each day on a continuous regimen for 2 years or until early termination from the study.
  Groups: 3
Drug: Placebo — There was no drug taken during study 3115A1-4000. During the 3115A1-303 study the test article was supplied as placebo capsules. Subjects took one capsule orally, once daily at approximately the same time each day on a continuous regimen for 2 years or until early termination from the study.
  Groups: 4

SUMMARY:
The objective of the study is to evaluate quantitative changes in mammographic breast density from baseline to 24 months in postmenopausal women receiving daily doses of either BZA 20 mg/CE 0.45 mg, BZA 20 mg/CE 0.625 mg, Raloxifene or placebo. The primary endpoint in this study is the change in mammographic breast density between baseline and month 24 for each group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed all scheduled evaluations in protocol 3115A1-303-WW.
* Completed 24 months of treatment in protocol 3115A1-303.
* Had a mammogram at the baseline visit and at the month 24 visit in protocol 3115A1-303, and both are original films that are technically acceptable for reading.
* Was at least 80% compliant with test article administration during protocol 3115A1-303.

Exclusion Criteria:

* Had a mammogram at either baseline or month 24 during the 3115A1-303 study that was technically unsatisfactory.
* One or both mammograms were digitized when they were obtained during the 3115A1-303 study.
* Had more than one mammogram at either the baseline or month 24 visit of study 3115A1-303.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with osteoporosis risk factors who were participants in a phase 3 trial for osteoporosis prevention (study 3115A1-303-WW)
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (22):
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Lousiville, Kentucky
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
- Pfizer Investigational Site, São Paulo, RS/Brazil, Brazil
- Pfizer Investigational Site, Nijmegen, Netherlands
- Norway (2):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Hamar

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3115A1-4000&StudyName=Study%20Evaluating%20Changes%20In%20Mammographic%20Breast%20Density

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had received bazedoxifene 20 milligram (mg)/conjugated estrogen 0.45 mg, bazedoxifene 20 mg/conjugated estrogen 0.625 mg, raloxifene 60 mg, or placebo in the primary study 3115A1-303 (NCT00675688) for up to 2 years and met the eligibility criteria were eligible to enroll in this study.
Groups:
- Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg: Participants who received bazedoxifene 20 mg/conjugated estrogen 0.45 mg tablet-in-capsule orally once daily at approximately the same time each day continuously for 24 months in the primary study 3115A1-303 (NCT00675688), provided mammograms at primary study baseline and Month 24 for digitization and subsequent analysis in this study.
- Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg: Participants who received bazedoxifene 20 mg/conjugated estrogen 0.625 mg tablet-in-capsule orally once daily at approximately the same time each day continuously for 24 months in the primary study 3115A1-303 (NCT00675688), provided mammograms at primary study baseline and Month 24 for digitization and subsequent analysis in this study.
- Raloxifene 60 mg: Participants who received raloxifene 60 mg tablet-in-capsule orally once daily at approximately the same time each day continuously for 24 months in the primary study 3115A1-303 (NCT00675688), provided mammograms at primary study baseline and Month 24 for digitization and subsequent analysis in this study.
- Placebo: Participants who received placebo capsule orally once daily at approximately the same time each day continuously for 24 months in the primary study 3115A1-303 (NCT00675688), provided mammograms at primary study baseline and Month 24 for digitization and subsequent analysis in this study.
Period: Overall Study
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Raloxifene 60 mg | Placebo
Started | 132 | 111 | 129 | 135
Completed | 132 | 111 | 129 | 135
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Raloxifene 60 mg | Placebo | Total
Number analyzed (Participants) | 132 | 111 | 129 | 135 | 507
Age, Customized [Number; unit: participants]
  Less than 50 years | 20 | 19 | 14 | 24 | 77
  50 to 65 years | 105 | 84 | 101 | 96 | 386
  Greater than or equal to 65 years | 7 | 8 | 14 | 15 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 111 | 129 | 135 | 507
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mammographic Breast Density at Month 24
Description: The digitized mammogram pairs were analyzed by a single trained radiologist who determined the density of the breast using software. The only left craniocaudal view was used for assessing breast density.
Time Frame: primary study baseline, Month 24
Population: All available participants were analyzed. Here, 'N' (number of participants analyzed) signifies those participants who had technically acceptable mammograms available at primary study baseline and Month 24.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Raloxifene 60 mg | Placebo
Number analyzed (Participants) | 129 | 105 | 125 | 126
percent change | -0.39 (1.75) | -0.05 (1.68) | -0.23 (1.76) | -0.42 (1.72)

ADVERSE EVENTS:
Description: This study was not designed to evaluate safety, because safety was evaluated in the primary study 3115A1-303 (NCT00675688). No safety data were collected and reported in this retrospective observational study.
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Raloxifene 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.